CLINICAL TRIAL: NCT01386762
Title: Effect of Intense Multi-modal Training on Bone Health and Quality of Life in Persons With Spinal Cord Injury
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: California State University, San Marcos (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Todd A. Astorino Ph.D, CSU--San Marcos
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 85756
Record Dates: First submitted 2011-06-30; First posted 2011-07-01 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Spinal Cord Injury; Obesity
Keywords: paralysis; paraplegia; obesity
MeSH Terms: conditions — Spinal Cord Injuries; Obesity; Paralysis; Paraplegia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise intervention (Experimental): 6 months of intense multimodal training.
  Interventions: Other: Exercise training

INTERVENTIONS:
Other: Exercise training — 6 months of intense multi-modal exercise consisting of vibration exercise, gait training, electrical stimulation, etc.

SUMMARY:
Bone loss is a common secondary complication of spinal cord injury (SCI), and treatments used to reverse this condition have equivocal effectiveness. The aim of this study is to determine the effect of intense multi-modal training on bone health, body fat, and quality of life in persons with SCI. Participants will complete 6 months of training during which various measures will be obtained at 0, 3, and 6 months. Control subjects are also being recruited to complete testing but not participate in training.

ELIGIBILITY:
Inclusion Criteria:

* Stable spinal cord injury below C2
* doctor's permission to participate in the study
* non-pregnant

Exclusion Criteria:

* see above

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-06; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density | 6 months
  Bone mineral density of the total body, knee, hip, and spine will be assessed via dual energy x-ray absorptiometry.

SECONDARY OUTCOMES:
Body fat | 6 months
  Total-body and regional depots of fat and fat-free mass will also be assessed in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- CSU--San Marcos Human Performance Lab, San Marcos, California, United States